CLINICAL TRIAL: NCT03527056
Title: Pilot Study Using Oral Capsule Fecal Microbiota Transplant To Decolonize Gastrointestinal Carbapenem-Resistant Enterobacteriaceae (CRE)
Brief Title: Pilot Study Using Oral Capsule FMT to Decolonize GI CRE
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: University of California, Los Angeles (Other)
Collaborators: OpenBiome (Industry); Finch Research and Development LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001946
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Enterobacteriaceae Infections; Fecal Microbiota Transplantation
Keywords: CRE
MeSH Terms: conditions — Enterobacteriaceae Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral capsule fecal transplantation (Experimental): Enrolled patients who have screened positive for CRE in the stool will receive fecal transplant via OpenBiome oral capsules. The patient is given 90 minutes to swallow all capsules and does not require any anesthesia or sedation. Stool samples to test for CRE will be taken 10 days and 30 days after the fecal transplant.
  Interventions: Biological: Fecal Microbiota Transplantation
- Observation (No Intervention): Enrolled patients who have screened positive for CRE in the stool will have stool samples to test for CRE taken 10 days and 30 days after initial enrollment.

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — This is a parallel arm study. All participants in the experimental arm will receive a single fecal transplantation via oral capsules to determine effectiveness and safety in decolonizing gastrointestinal CRE.
  Other Names: FMT; Fecal Transplant
  Arms: Oral capsule fecal transplantation

SUMMARY:
Carbapenem-Resistant Enterobacteriaceae (CRE) are bacteria that have become resistant to carbapenems by producing enzymes that break down carbapenems. The prevalence of CRE continues to rise globally but the treatment options are extremely limited. In case series, isolation of CRE from any site, whether there is clinical infection or not, has been associated with all-cause hospital mortality ranging from 29% to 52%. There are no known methods for reliably decolonizing gastrointestinal (GI) CRE. In rare case reports, fecal microbiota transplant (FMT) has successfully eradicated gastrointestinal colonization of CRE, but there has been no larger study further investigating this. FMT via oral capsules is the least invasive method and has demonstrated efficacy and short-term safety in treating patients with recurrent Clostridium difficile infections. Therefore, the investigators propose this pilot study to determine the effectiveness of oral capsule fecal transplantation in the decolonization of gastrointestinal CRE.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Have intestinal carriage of CRE

Exclusion Criteria:

* Pregnant
* Peripheral WBC >12 x 10^9/L and/or temperature >38 degrees Celsius
* Swallowing dysfunction or known chronic aspiration
* Delayed gastric emptying
* History of intestinal obstruction
* Active CRE infection
* Acute exacerbation of underlying comorbid condition
* Severely immunocompromised patients
* Inflammatory bowel disease
* Allergies to ingredients Generally Recognized as Safe
* Adverse event attributable to previous FMT
* Concomitant antibiotic use or antibiotic use 48 hours before FMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with CRE decolonization at day 10 (+/- 3 days) after fecal transplant | 10 days
  CRE decolonization is defined by absence of CRE on stool culture using standard clinical laboratory techniques. Stool samples will be collected 10 days after FMT.
Proportion of participants with an adverse event through day 10 (+/- 3 days) after FMT | 10 days
  Telephone calls are made to participants 10 days after FMT to assess for adverse event, severe adverse event, and adverse events of special interest (newly acquired transmissible infectious diseases).

SECONDARY OUTCOMES:
Proportion of participants with CRE decolonization at month 1 (+/-5 days) after FMT | 1 month
  CRE decolonization is defined by absence of CRE on stool culture using standard clinical laboratory techniques. Stool samples will be collected 30 days after FMT.
Proportion of participants with CRE infection at day 10 (+/-3 days) and month 1 (+/-5 days) after FMT | 1 month
  CRE infection will be defined as an associated bacteremia, urinary tract infection, wound-related infection or other clinical infection deemed to be CRE associated at the discretion of the treating physician.
Proportion of participants with an adverse event, severe adverse event, or adverse events of special interest through month 1 (+/-5 days) after FMT. | 1 month
  Telephone calls are made to participants 1 month after FMT to assess for adverse event, severe adverse event, and adverse events of special interest (newly acquired transmissible infectious diseases).
Proportion of participants with a severe adverse event at month 6 (+/-14 days) after FMT. | 6 months
  Telephone calls are made to participants 6 months after FMT to assess for severe adverse event.
Proportion of participants with microbial engraftment assessed by microbiome disruption index (MDI) (MDI-community and MDI-species) measured by 16s ribosomal RNA at time of enrollment, day 10 (+/-3 days) and month 1 (+/-5 days) after FMT | 1 month
  Stool samples collected at baseline before FMT, day 10 after FMT, 1 month after FMT will be sent for 16s sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rubin, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No